CLINICAL TRIAL: NCT06290531
Title: Different Methods for Reducing Buccal Infiltration Local Anesthesia Injection Pain in Children: A Randomized Controlled Study.
Brief Title: Different Methods for Reducing Buccal Infiltration Local Anesthesia Injection Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Abdelgawad, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CEBD-CU-2023-11-12
Record Dates: First submitted 2024-01-29; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Dental Caries in Children
Keywords: Local Anesthesia; Buzzy; Topical Anesthesia; Pain; precooling
MeSH Terms: conditions — Pain

STUDY DESIGN:
Masking Description: The statistician was only blinded for data analysis. But it was not feasible to blind the participant, investigator or the outcome assessor due to the nature of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Buzzy device (cold and vibration) (Experimental)
  Interventions: Device: Buzzy device (cold and vibration)
- Buzzy device (vibration only) (Experimental)
  Interventions: Device: Buzzy device (vibration only)
- Precooling (Experimental)
  Interventions: Other: precooling
- Flavored Benzocaine topical anesthetic gel 20% (Active Comparator)
  Interventions: Other: Flavored Benzocaine topical anesthetic gel 20%

INTERVENTIONS:
Device: Buzzy device (cold and vibration) — The device produces cold and vibration to act on the gate control theory and provide painless injection by nerve distraction
  Arms: Buzzy device (cold and vibration)
Device: Buzzy device (vibration only) — The device produces vibration to act on the gate control theory and provide painless injection by nerve distraction
  Arms: Buzzy device (vibration only)
Other: precooling — Ice cubes used for applying coolness at the injection area
  Arms: Precooling
Other: Flavored Benzocaine topical anesthetic gel 20% — Topical anesthetic gel
  Arms: Flavored Benzocaine topical anesthetic gel 20%

SUMMARY:
Local anesthetic injection is considered one of the most annoying dental procedures. The use of topical anesthesia is considered a routine procedure in the dental clinic especially for children. However, the taste and application procedure of the topical gel may not be pleasant for all children.

The introduction of the Buzzy device is considered a distraction measure in the medical field. Alanazi et al., 2019, studied the effect of using the Buzzy device with cold and vibration compared to the conventional infiltration technique using 30-gauge needle. They concluded that the use of the Buzzy device resulted in better patients' acceptance and significantly lower Wong-Baker scores.

Ballard et al., 2019, mentioned in their systematic review the efficacy of the Buzzy device for pain management during needle-related procedures, they concluded that the use of the device may be promising. Ghaderi et al., 2013, evaluated the effect of cooling the injection site on pain perception before infiltration of local anesthetics. They found that cooling the injection site before infiltration of local anesthetics in the buccal mucosa for 1 min, reduced pain perceived by pediatric patients.

DETAILED DESCRIPTION:
The investigators used the topical anesthesia, Buzzy device (using vibration only and using cold and vibration) or precooling on pain during buccal infiltration local anesthesia injection.

ELIGIBILITY:
Inclusion Criteria:

* Children in the mixed dentition stage,
* Age range 6-12 years old,
* Need extraction to a maxillary molar,
* Cooperative and medically free.

Exclusion Criteria:

* Exclusion will be performed if the parent refused the participation of their children in the research.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2022-01-16 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Patient reported pain during needle injection | Immediately post injection
  Patient was asked to choose from the faces on the Wong Baker faces pain rating scale (0-10) with 10 is the worst score

SECONDARY OUTCOMES:
Child behaviour during needle injection | Immediately during injection
  Child behaviour during needle injection was recorded using Sound-eye-motor scale (0-9) with 9 is the worst score
Heart rate | Immediately post injection
  Heart rate was recorded using pulse oximetry (beats/minute)
Oxygen saturation | Immediately post injection
  Oxygen saturation was recorded using pulse oximetry
Child and parent satisfaction | Immediately post injection
  By asking questions to both child and their parent on a likert scale for children ( positive, neutral and negative) for parents ( strongly agree, agree, no opinion, disagree and strongly disagree)

CONTACTS AND LOCATIONS:
Overall Officials: Fatma KI Abdelgawad, PhD, Principal Investigator — Associate Professor
Locations (1):
- Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No